CLINICAL TRIAL: NCT00683644
Title: Zinc to Treat Tinnitus in the Elderly: A Randomized Placebo Controlled Crossover Trial.
Brief Title: Zinc to Treat Tinnitus in the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Tinnitus Research Initiative (Other)
Responsible Party: Principal Investigator, Richard Tyler, Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200603807
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Tinnitus
Keywords: tinnitus, zinc
MeSH Terms: conditions — Tinnitus | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: placebo pill
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 - zinc placebo (Experimental): Zinc sulfate (50 mg elemental zinc) taken once daily for 4 months. Washout 1 month. Placebo oral capsule taken once a day for 4 months.
  Interventions: Drug: Zinc; Drug: Placebo oral capsule
- 2 - placebo zinc (Experimental): Placebo oral capsule taken once a day for 4 months. Washout 1 month. Zinc sulfate (50 mg elemental zinc) taken once daily for 4 months.
  Interventions: Drug: Zinc; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Zinc — Zinc taken once daily
  Other Names: zinc sulfate
Drug: Placebo oral capsule — Placebo capsules taken once daily
  Other Names: Placebo

SUMMARY:
There is widespread belief and some evidence to indicate that zinc can successfully treat tinnitus. Zinc deficiency is more likely to occur in the elderly . The primary objective of this study is to establish the effectiveness of zinc for the treatment of tinnitus in individuals 60 years of age and older. Subjects will be randomly assigned to either receive zinc daily or a placebo. After 4 months and a 1-month wash-out, the subjects will be crossed over to the other group.

DETAILED DESCRIPTION:
There is widespread belief and some evidence to indicate that zinc can successfully treat tinnitus. Zinc deficiency is more likely to occur in the elderly . The primary objective of this study is to establish the effectiveness of zinc for the treatment of tinnitus in individuals 60 years of age and older. Subjects will be randomly assigned to either receive zinc daily or a placebo. After 4 months and a 1-month wash-out, the subjects will be crossed over to the other group. 116 patients were tested. Tinnitus loudness and the Tinnitus Handicap Questionnaire are the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Tinnitus for 6 months or more
* Normal copper levels
* Be generally healthy

Exclusion Criteria:

* Have a treatable otological disorder
* Involved in litigation
* Have or are suspected of having a serious psychiatric problem
* Involved in other treatments for tinnitus
* Are taking drugs which might interact with zinc and result in tinnitus
* Have copper deficiency
* Have Zinc levels above normal
* Are cognitively impaired.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Tyler, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coelho C, Witt SA, Ji H, Hansen MR, Gantz B, Tyler R. Zinc to treat tinnitus in the elderly: a randomized placebo controlled crossover trial. Otol Neurotol. 2013 Aug;34(6):1146-54. doi: 10.1097/MAO.0b013e31827e609e. PMID 23598691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited from audiology clinic in otolaryngology department
Groups:
- Group 1 Zinc First: Zinc sulfate (50 mg elemental zinc) taken once daily for 4 months ZINC 4 MONTHS WASHOUT 1 MONTH PLACEBO 4 MONTHS
- Group 2 Placebo First: Placebo capsules taken once a day for 4 months
  PLACEBO 4 MONTHS WASHOUT 1 MONTH ZINC 4 MONTHS
Period: Overall Study
Arm/Group | Group 1 Zinc First | Group 2 Placebo First
Started | 58 | 58
Completed | 45 | 44
Not Completed | 13 | 14
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Low copper, other health problems, | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Zinc First: Zinc sulfate 220 mg capsules, (corresponding to 50 mg of elemental zinc) administered once a day for 4 months. Washout period of 30 days. Placebo capsules administered once a day for 4 months.
- Group 2 Placebo First: Placebo capsules administered once a day for 4 months. Washout period of 30 days. Zinc sulfate 220 mg capsules, (corresponding to 50 mg of elemental zinc) administered once a day for 4 months.
- Total: Total of all reporting groups
Arm/Group | Group 1 Zinc First | Group 2 Placebo First | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (5.5) | 67.8 (5.8) | 67.8 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 34 | 38 | 72
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 109
Tinnitus Handicap Questionaire [Mean (Standard Deviation); unit: units on a scale] | 28.4 (20.3) | 27.4 (19.2) | 27.9 (19.8)
Tinnitus Annoyance Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Tinnitus annoyance rate on a scale of 0 (no annoyance) to 100 (maximum degree of annoyance)
  units on a scale | 60 (22.7) | 65.8 (23) | 63 (23.1)
Tinnitus Loudness Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Tinnitus loudness rate on a scale of 0 (no perception of tinnitus) to 100 (highest degree of tinnitus perception)
  units on a scale | 66.7 (16.2) | 67.5 (15.1) | 67.3 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tinnitus Reaction on the Tinnitus Handicap Questionnaire Scores (0-100) at 4 Months
Description: Validated questionnaire of tinnitus reactions. Scale 0 (no tinnitus reaction)- 100 (worst tinnitus reaction). Our primary outcome was the difference scores between Tinnitus Handicap Questionnaire (THQ) on baseline and end of treatment on zinc and placebo treatment. As stated by Newman et al., the test-retest variability was 20%, and difference scores greater than this should be considered a significant reduction. Therefore, changes on the difference scores of 20 or greater were considered as a statistically significant and therefore clinically meaningful improvement for THQ. The minimum score is zero and the maximum is 100. 0 is better and 100 is worse. This applies to all outcome measures.
Time Frame: baseline - 4 months
Population: For data analysis purposes subjects were recombined in 2 groups (Zinc and Placebo). Group ZINC: subjects who completed 4 months with Zinc 50 mg daily either from baseline to month 4, or after washout (from month 5 to 9). Group PLACEBO: subjects who completed 4 months with placebo either from baseline to month 4, or after washout (from month 5 to 9)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Zinc: Participants that completed 4 months taking Zinc (50 mg) daily, either from baseline to month 4, or after washout period, from month 5 to 9).
- Placebo: Participants that completed 4 months taking placebo capsules daily, either from baseline to month 4 or after a washout period of 1 month (from month 5 to month 9).
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 93 | 94
units on a scale
  THQ scores at Baseline | 22.03 (22) | 24.9 (20.7)
  THQ scores at 4 months | 23.7 (18.7) | 25.4 (21.3)
Statistical Analysis 1: Comparison: Zinc vs Placebo; Test type: Other — The observed power in THQ for zinc is 0.16, and that for placebo is 0.06; p > 0.05, Chi-squared — Threshold for significance is 0.05

2. Secondary Outcome: Changes on Baseline Tinnitus Magnitude on Tinnitus Loudness Rating Scores (0-100) at 4 Months Treatment
Description: Participants should rate their tinnitus loudness on a scale of 0 (no perception of tinnitus) to 100 (highest degree of tinnitus perception).
Time Frame: baseline and 4 months
Population: Subjects that complete 4 months treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Zinc: Participants who completed 4 months taking Zinc (50 mg) daily, either from baseline to month 4, or after washout period, from month 5 to 9).
- Placebo: Participants who completed 4 months taking placebo capsules daily, either from baseline to month 4, or after washout period of 1 month (from month 5 to 9).
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 93 | 93
units on a scale
  Baseline tinnitus loudness rating scores (SD) | 67.7 (18.7) | 66 (18.4)
  4 months tinnitus loudness rating scores (SD) | 68.1 (21.4) | 67.6 (20.2)
Statistical Analysis 1: Comparison: Zinc; Test type: Other; p = 0.89, paired t test — Threshold for significance is 0.05
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.36, paired t test — Threshold for significance is 0.05

3. Secondary Outcome: Changes on Baseline Tinnitus Reactions on Tinnitus Annoyance Rating Scores (0-100) at 4 Months Treatment
Description: Tinnitus annoyance rate on a scale of 0 (no annoyance) to 100 (maximum degree of annoyance)
Time Frame: baseline and 4 months
Population: Subjects that complete 4 months treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Zinc: Zinc sulfate: Zinc sulfate capsules corresponding to 50 mg of elemental zinc, taken once daily. Period of use: 4 months, either on baseline or month 5 (after a washout period: 1 month)
- Placebo: Placebo taken once daily. Period of use: 4 months, either on baseline or month 5 (after a washout period of 1 month)
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 93 | 93
units on a scale
  Baseline tinnitus annoyance rating scores | 59.67 (25.40) | 57.7 (30.85)
  4 months tinnitus annoyance rating scores | 61 (30.5) | 57.9 (26.7)
Statistical Analysis 1: Comparison: Zinc; Test type: Other; p = 0.64, paired t test — Threshold for significance is 0.05
Statistical Analysis 2: Comparison: Placebo; Test type: Other; p = 0.93, paired t test — Threshold for significance is 0.05

ADVERSE EVENTS:
Time Frame: 9 months
Description: There were 99 participants at risk while receiving Zinc and 101 participants at risk when receiving Placebo.
Groups:
- Zinc: 54 participants received Zinc first and 45 participants received Zinc after 1 month washout. The total number of participants at risk to Zinc is 99.
- Placebo: 55 participants received Placebo first and 46 participants received Placebo after 1 month washout. The total number of participants at risk to Placebo is 101.
Arm/Group | Zinc | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/101
Other Adverse Events (participants affected / at risk) | 1/99 | 2/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc (N=99) | Placebo (N=101)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metallic taste (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
For data analysis purposes subjects were divided "per intervention". Zinc: subjects who completed 4 mo with zinc from baseline to month 4, or after washout. Placebo: subjects who completed 4 mo with placebo from baseline to month 4, or after washout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No